CLINICAL TRIAL: NCT02108366
Title: A Randomized Controlled Trial on the Treatment of Severe Influenza A Infection
Brief Title: Treatment of Severe Influenza A Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Ivan FN Hung, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 13-009
Record Dates: First submitted 2014-03-31; First posted 2014-04-09 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Influenza, Human
Keywords: severe; influenza A; celecoxib
MeSH Terms: conditions — Influenza, Human; Lymphoma, Follicular | interventions — Celecoxib; Oseltamivir; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo + oseltamivir 75mg bid for 5 days
  Interventions: Drug: Oseltamivir; Drug: Placebo
- Celecoxib (Experimental): Celecoxib 200mg daily + oseltamivir 75mg bid for 5 days
  Interventions: Drug: Celecoxib; Drug: Oseltamivir

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 200mg daily
  Other Names: COX II inhibitor
  Arms: Celecoxib
Drug: Oseltamivir — Oseltamivir 75mg bid
  Other Names: Tamiflu
Drug: Placebo — Placebo capsule identical in appearance to celecoxib capsule, containing corn starch
  Other Names: Corn starch
  Arms: Placebo

SUMMARY:
Each year, influenza A infection caused great mortality and morbidity, especially among the elderly and individuals with chronic illness. Many of these patients are 'late presenters' who are admitted to hospital a few days after symptoms onset and have developed complications secondary to immunodysregulation. Antiviral treatment with the neuraminidase inhibitor is of limited usage for patients who presented to the hospital 48 hours after symptom onset. Apart from ventilatory and extracorporeal membrane oxygenation support, treatment options for these patients are limited. Recent animal study has demonstrated that combinations of an antiviral agent with a COX-II inhibitor can reduce mortality in mice infected with influenza virus. The investigators therefore propose to enrol patients with severe influenza A infection requiring hospitalization and oxygen support on a randomized controlled trial with celecoxib.

DETAILED DESCRIPTION:
The aim of this double blind randomized controlled trial is to compare the clinical efficacy and safety of celecoxib combined with neuraminidase inhibitors in patients with severe influenza A infection. The hypothesis of this study is that treatment of severe influenza A infection with celecoxib will reduce mortality. The primary outcome to be assessed will be the 28-days mortality rate from hospitalization. The secondary outcomes to be assessed will be safety of the treatment, duration of intensive care, duration of ventilatory and oxygen support, the viral load and cytokine change.

ELIGIBILITY:
Inclusion Criteria:

1) Male or female patients ≥18 years 2) Written informed consent by patient or next-of kin (if patient is too ill to consent) 3) Presumptive diagnosis of influenza A satisfying both clinical and laboratory criteria. The laboratory criteria are defined as at least one RT-PCR positive for influenza A (H1N1, H3N2, H5N1 and H7N9) from respiratory clinical specimens including nasopharyngeal samples and endotracheal aspirates. The clinical criteria are defined as hospitalization with fever or one of the symptoms suggestive of influenza infection including sore throat, rhinorrhea, cough or shortness of breath 2) Desaturation to <90% in room air by pulse oximetry and required oxygen supplement 3) Within 7 days of onset of symptoms. Patients have to fulfil all the aforementioned criteria.

Exclusion Criteria:

1) Age <18 years. 2) A known hypersensitivity to celecoxib, oseltamivir or zanamivir 3) Unable to obtain informed consents 4) Influenza A infection diagnosed beyond 7 days from symptom onset 5) Patients receiving other antiviral treatment (apart from oseltamivir or zanamivir), N-acetylcystiene, statins and tradition Chinese medicine during the current admission 6) Patients with renal impairment of creatinine clearance < 30mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 28 days
  28 days mortality from hospitalization

SECONDARY OUTCOMES:
Viral load | 7 days
  1 day before treatment for 1 week
Cytokine | 7 days
  1 day before treatment for 7 days
Intensive care stay | An expected average of 2 weeks
  Period under intensive care
Ventilatory support period | An expected average of 2 weeks
  Duration of patient on ventilatory support
Systemic adverse events | 1 week
  from commencement of treatment for 1 week
Hospitalization | An expected average of 4 weeks
  from hospital admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN HUNG, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- Ivan Hung, Hong Kong, Hong Kong